CLINICAL TRIAL: NCT03776214
Title: LYMPHOSPIR : Impact of Surgery in Addition to Optimal Management of Lymphedema.
Brief Title: Surgery in Addition to the Medical Treatment of Lymphedema
Acronym: LYMPHOSPIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Department of Reconstructive surgery, UH Montpellier (Unknown); Department of vascular medecine, UH Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0133
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Optimal Treatment of Lymphedema
Keywords: No pitting edema; After medical and surgical evaluation; Microlipoaspiration; surgery; lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphedema is a chronic pathology with a real impact on the quality of life of patients. Despite optimal medical management of patients, some patients still have no pitting edema on which the medical treatment has no effect.

It is adipose tissue secondary to the evolution of lymphedema. It is often painful and important in terms of volume with the resulting functional consequences. The investigators propose to these patients a surgical management complementary to the optimal medical treatment by microlipoaspiration associated or not with a dermolipectomy. This surgical management began in 2014 in our service. The investigators want to evaluate the impact on quality of life of patients in this surgical management in addition to medical care.

DETAILED DESCRIPTION:
Detailed Description:

This is a monocentric, observational cohort study.

Main judgment criteria:

Evolution of the quality of life score of the LYMQOL self-questionnaire between preoperative and postoperative (at 3.6 and 12 months) The investigators used a French translation of Keeley's LYMQOL (Quality Of Life Measure for Limb Lymphoedema) self-administered questionnaire in 2010 (2) to assess the quality of life of patients. This is a lymphedema specific questionnaire for which there is one version for the upper limb and one for the lower limb. Limb function, lymphedema symptoms, body image and mood are assessed independently. It allows to obtain a score between 1 and 4 which corresponds to the discomfort felt. The higher the score, the better the quality of life. It also includes, in the last question, a numerical scale allowing the patient to note her quality of life between 0 and 10.

Since 2016, patients have systematically completed quality of life questionnaires. Perimeter measurements are also done systematically at each visit, these data are available in the patient's computerized medical records (Dx Care).

Secondary judgment criterion:

Difference in the volume of the limb operated between preoperative and postoperative (3, 6 and 12 months)

The volume is calculated on the basis of stepped circumferential measurements (every 10 cm starting from the patella for the lower limb and every 5 cm starting from the bend of the elbow for the upper limb). These measures are taken at each consultation by our physiotherapists, specialized nurses or vascular doctors.

It is therefore a question of retrospectively analyzing the data collected.

The data will then be anonymised by a two-letter code and a number and will be entered on a Excel file available on a secure directory of the CHU for analysis.

A dedicated support protocol is already implemented in the Cf Appendix service. There are no special modalities for patients not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* no pitting edema
* good therapeutic compliance
* weight stability

Exclusion Criteria:

- under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with lymphedema (primary or secondary) of arm or limb selected by the medical and chirurgical staff (no pitting edema, optimal medical treatment, good therapeutic compliance) for an liposuccion or dermolipectomia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
quality of life (self questionnaire LYMQOL) | 1 day
  To evaluate the impact of surgery in addition to the medical management of lymphedema on the quality of life of operated patients between preoperative and postoperative

SECONDARY OUTCOMES:
volume of operated limb | 1 day
  Evaluate the effectiveness of surgery in addition to medical management in terms of volume reduction of the operated limb between preoperative and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: MESTRE GODIN Sandrine, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC